CLINICAL TRIAL: NCT06067204
Title: Prehospital Automatic Ventilation on Resuscitation Outcomes in Out-of-hospital Cardiac Arrest Patients: a Randomized Controlled Trial
Brief Title: Automatic Ventilation in Prehospital Resuscitation on OHCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202304132RINB
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: automatic ventilation; prehospital resuscitation; emergency medical service
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the emergency medical service crew will know the intervention in each participant. The patient will not be aware of the type of ventilation strategy because of OHCA status. The investigator and outcomes assessor will not able to acquire the allocation results until the study ends.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Automatic ventilation (Experimental): After the advanced airway is placed, an automatic pneumatic ventilator will be connected and provides ventilation in every 6 seconds.
  Interventions: Device: Automatic ventilation
- Manual ventilation (Active Comparator): After the advanced airway is placed, a bag valve mask resuscitator will be connected and provides ventilation in every 6 seconds by the emergency medical technician.
  Interventions: Device: Manual ventilation

INTERVENTIONS:
Device: Automatic ventilation — The FDA-approved device used is "Meditech" MICROVENT RESUSCITATOR, which is connected to the endotracheal tube, supraglottic airway or tracheostomy tube. It is powered by the airflow from the oxygen tank and provides ventilation in fixed interval. It has a pressure valve which will release the pressure once the airway pressure exceeds its threshold. In the current study, the threshold is set at 60 mmH2O. The tidal volume is set at 500-600 ml.
  Other Names: automatic pneumatic ventilation (APV)
  Arms: Automatic ventilation
Device: Manual ventilation — The adult size bag-valve mask is connected to the endotracheal tube, supraglottic airway or tracheostomy tube. The interval, pressure and volume of the ventilation is controlled by the emergency medical technicians.
  Other Names: Bag-valve-mask (BVM) ventilation
  Arms: Manual ventilation

SUMMARY:
The goal of this randomized controlled trial is to compare prehospital ventilation strategies in out-of-hospital cardiac arrest. The intervention group is automatic ventilation and the control group is manual ventilation. The main questions it aims to answer are:

1. How does automatic ventilation affect OHCA patients' survival and prognosis comparing to manual ventilation.
2. What are the differences on resuscitation qualities between automatic ventilation and manual ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old at the time of occurrence of out-of-hospital cardiac arrest (OHCA).
* Attended by the Hsinchu County Fire Department for emergency medical assistance.

Exclusion Criteria:

* Pregnant women.
* OHCA caused by trauma.
* Return of spontaneous circulation (ROSC) observed at the scene.
* Clearly deceased at the scene (reaching conditions such as decomposition, rigor mortis, severe burns, decapitation, evisceration, or trunk fracture).
* Refusal of medical transportation by family members.
* No placement of an advanced airway throughout the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of any return of spontaneous circulation (ROSC) | 2 hours
  The patient achieved ROSC in prehospital or inhospital resuscitation.

SECONDARY OUTCOMES:
The percentage of sustained ROSC in 24 hours | up to 24 hours
  The patient survives for 24 hours after arriving the hospital.
The percentage of survival to hospital discharge | up to 90 days
  The patient survives to discharge from the hospital.
The percentage of favorable neurological outcome after discharge | up to 90 days
  The patient survives to discharge from the hospital with Cerebral Performance Categories Scale 1 or 2.
Chest compression fraction | up to 1 hour
  The chest compression fraction during prehospital resuscitation recorded by the monitor.
The percentage of intravenous catheter placement | up to 1 hour
  Whether the patient has an IV catheter placed in the prehospital setting.
The percentage of epinephrine injection | up to 1 hour
  Whether the patient has epinephrine injected in the prehospital setting.
The satisfaction of emergency medical technician (EMT) during the dispatch | up to 5 hours
  The outcome contained five questions:
  * More convenient to use
  * Shorter time required to complete ventilation (from advanced airway placement to the start of ventilation)
  * Smoother patient transport process
  * Ability to perform more emergency medical techniques
  * Overall satisfaction with the execution of emergency medical tasks
  The EMTs answer in the 5-level scale (highly disagree, disagree, neutral, agree, highly agree)
The percentage of pneumothorax | up to 3 days
  Unilateral, bilateral or tension pneumothorax which might be associated with the ventilation strategy.

OTHER OUTCOMES:
Ventilation rate in the prehospital resuscitation | up to 1 hour
  The ventilation rate recorded by the portable monitor with feedback sensor (BVM help).
Tidal volume in the prehospital resuscitation | up to 1 hour
  The tidal volume recorded by the portable monitor with feedback sensor (BVM help).
Chest compression depth in the prehospital resuscitation | up to 1 hour
  The chest compression depth recorded by the portable monitor with feedback pad.
Chest compression rate in the prehospital resuscitation | up to 1 hour
  The chest compression rate recorded by the portable monitor with feedback pad.
End-tidal carbon dioxide level (ETCO2) | 1 hour
  The ETCO2 recorded in the prehospital resuscitation process.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Pei-Chuan Huang, M.D., M.S., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan CY, Huang SS, Chen CH, Sung CW, Chang CH, Hung TH, Liu YC, Huang EP. Prehospital ventilation strategies in out-of-hospital cardiac arrest: A protocol for a randomized controlled trial (PIVOT trial). Resusc Plus. 2024 Nov 16;20:100827. doi: 10.1016/j.resplu.2024.100827. eCollection 2024 Dec. PMID 39624188